CLINICAL TRIAL: NCT06565585
Title: Prediction of Local Recurrence and Its Impact on Long-term Outcomes After Low-risk Glans-sparing Surgery Defined as Wide Local Excision, Circumcision, Laser Ablation, Glans Resurfacing and Partial Glansectomy for Penile Squamous Cell Carcinoma
Brief Title: Prediction of Local Recurrence and Its Impact on Long-term Outcomes After Low-risk Glans-sparing Surgery for Penile Squamous Cell Carcinoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S66471
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Penile Cancer, Recurrent
Keywords: Penile cancer; Local recurrence; Organ-sparing surgery
MeSH Terms: conditions — Penile Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-risk Glans-sparing surgery patients: Patients with lower-risk tumors who underwent glans-sparing surgery defined as circumcision, wide local excision, laser ablation, glans resurfacing and partial glansectomy.
  Interventions: Procedure: Glans-sparing surgery
- High-risk glansectomy patients: Patients who underwent total glansectomy due to higher risk tumors resulting in a complete removal of all the glandulopreputhial epithelium.

INTERVENTIONS:
Procedure: Glans-sparing surgery — Patients who underwent glans-sparing surgery
  Groups: Low-risk Glans-sparing surgery patients

SUMMARY:
The treatment paradigm for primary penile squamous cell carcinoma (PSCC) has increasingly favored maximal organ preservation without compromising oncological outcomes. However, the literature has often included heterogeneous patient cohorts and varied surgical approaches, making it challenging to draw definitive conclusions about the impact of local recurrence (LR) on survival.

Since the investigators recently published the results from a large, multicentric international study on a homogeneous cohort of high-risk PSCC patients who were treated with upfront complete glansectomy, the investigators have been demonstrating that local recurrence after upfront glansectomy was strongly correlated with worse overall survival and cancer-specific survival in this more homogeneous cohort, therefore challenging the dogma that LR following organ-sparing surgery for PSCC does not affect survival outcomes (Roussel et al., BJU Int 2021; DOI: 10.1111/bju.15297).

The investigators hypothesized that these findings were caused by an enrichment of higher risk tumors in this cohort since solely glansectomy patients with a complete removal of all the glandulopreputhial epithelium were included. Consequently, the hypothesis has arisen that LR might not be a predictor of poorer survival outcomes in lower-risk tumors who underwent glans-sparing surgery defined as circumcision, wide local excision, laser ablation, glans resurfacing and partial glansectomy, and that previous findings influencing the guidelines may be heavily influenced by the inclusion of large proportions of low-risk tumors in rather heterogenous cohorts in terms of technical approach.

Therefore, this study aims to explore whether LR similarly affects survival in lower-risk tumors treated with glans-sparing techniques such as circumcision, wide local excision, glans resurfacing, laser ablation, and partial glansectomy.

DETAILED DESCRIPTION:
Penile squamous cell carcinoma (PSCC) is a rare disease with a limited body of evidence on which to base management decisions. The World Health Organization (WHO) has estimated 36,068 new cases of penile cancer in 2020, with an age-standardized incidence of 0.8 per 100,000 people worldwide. Traditionally performed partial or total penectomy have been associated with significant comorbidity with respect to altered voiding, sexual function, appearance, and psychological well-being.

In terms of treatment of the primary the European Association of Urology (EAU) guidelines recommend performing complete tumor removal with as much organ preservation as possible, without compromising oncological control. Organ-sparing surgery (OSS) encompasses a plethora of surgical techniques including wide local excision, circumcision, glans resurfacing, and partial or total glansectomy.

Consequently, penile-sparing approaches have been increasingly employed, with excellent functional outcomes and significant improvements in patients' quality of life compared to radical treatment. This trend towards OSS is based on the fact that, although patients treated with penile preservation experience more local recurrence (LR) compared to partial or total penectomy, the occurrence of LR did not compromise survival in several previously studied cohorts with a heterogeneous patient population including both high-risk and low-risk tumors.

However, the investigators recently published the results from a large, multicentric international study on a homogeneous cohort of high-risk patients who were treated with upfront complete glansectomy. It was found that LR after upfront glansectomy represents an underlying aggressive disease course and was strongly correlated with worse overall survival (HR 2.89, 95% CI 2.02-4.14, <0.001) and cancer-specific survival (HR 5.64, 95% CI 3.45-9.22, P < 0.001) in this cohort, therefore challenging the dogma that LR following OSS for PSCC does not affect survival outcomes. Multivariable Cox proportional hazards regression analysis identified pT3 stage and high-grade disease as independent predictors of LR.

The investigators hypothesized that these findings were caused by an enrichment of higher risk tumors in our cohort, since solely glansectomy patients who undergo a complete removal of all the glandulopreputhial epithelium were studied. Conversely, the investigators would hypothesize that LR might not be a predictor of poorer survival outcomes in lower risk tumors who undergo wide local excision, partial glansectomy, laser ablation, circumcision or glans resurfacing. This would be the reason that previous, heterogenous cohorts, including these techniques did not find an adverse effect of LR on survival outcomes.

Therefore, the aim of this study is to study predictive pathological factors for LR as well as the impact of LR on long-term survival outcomes solely in patients who are treated with wide local excision, partial glansectomy, laser ablation, circumcision and glans resurfacing, reflecting a lower risk OSS patient population, defined as glans-sparing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Underwent low-risk OSS defined as: wide local excision, partial glansectomy, laser ablation, circumcision, and glans resurfacing for PSCC

Exclusion Criteria:

* Underwent partial or total penectomy as primary surgery
* regional lymph node involvement at presentation (cN+ stage)
* metastates at presentation (cM+ stage)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will collect data from patients operated in high-volume penile cancer centers on in the period from 1st of January 2000 to 1st of June 2023. All patients should have undergone glans-sparing surgery.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
long-term oncologic outcomes (OS, CSS) | 1/01/2000 - 1/06/2023
  impact of local recurrence after glans-sparing surgery on long-term oncologic outcomes (OS, CSS)

SECONDARY OUTCOMES:
Predictive histopathological factors for local recurrence | 1/01/2000 - 1/06/2023
  Identify histopathological factors that might predict the occurrence of local recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Albersen, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No